CLINICAL TRIAL: NCT00059111
Title: Mechanisms Mediating Cardiovascular Disease in Children With Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1212; R01HL070907-01A1 (NIH)
Record Dates: First submitted 2003-04-17; First posted 2003-04-18 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Sleep Apnea Syndromes; Lung Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Sleep Apnea Syndromes; Lung Diseases; Hypertension

SUMMARY:
To identify the early effects of obstructive sleep apnea on the cardiovascular system of children.

DETAILED DESCRIPTION:
BACKGROUND:

Obstructive sleep apnea (OSA) is an important clinical disorder occurring in men, women, and children with a prevalence of 4 percent, 2 percent and 1-3 percent, respectively. OSA is under active study in adults and is definitely linked with increased cardiovascular morbidity, even in its mild to moderate clinical forms. In contrast, OSA has not been well studied in children and the potential deleterious consequences on cardiovascular function have received little or no attention.

DESIGN NARRATIVE:

The study will examine in children 1) The interaction between OSA and baroreflex dysfunction, 2) The relation of OSA severity and baroreflex dysfunction to abnormalities in blood pressure control during wakefulness and sleep, 3) The association of the diminished baroreflex gain and impaired blood pressure control with an index of end organ damage, the left ventricular mass index, and 4) Whether effective treatment of OSA results in significant improvement in baroreceptor function, blood pressure control and a decrease in left ventricular mass index. A cross-sectional study will be conducted in 8-12 year old children with OSA and a matched group of normal children. Studies include baroreceptor function, 24-hour ambulatory blood pressure and left ventricular mass index. Baroreceptor function will be measured by non-invasive techniques based on combined computer analysis of heart rate and blood pressure measured by portapres. 24-hour ambulatory blood pressure will be measured by a Spacelab monitor and left ventricular mass index will be measured by direct M-mode echocardiogram. A longitudinal study will be conducted on the effect of adequate treatment of OSA on baroreceptor function, daytime and nocturnal blood pressure and left ventricular mass index. A cohort of children with OSA and a matched group of normal controls will be followed for a period of 12 months after treatment of the disorder. Results are expected to show that children with OSA have decreased baroreceptor sensitivity, elevated nocturnal blood pressure and increased left ventricular mass index and that effective therapy for OSA, as determined by polysomnography, will improve or normalize baroreceptor sensitivity as well as nocturnal blood pressures and will lead to a decrease in left ventricular mass index.

ELIGIBILITY:
No eligibility criteria

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raouf Amin — Children's Hospital & Medical Center

REFERENCES:
- [Background] Amin RS, Kimball TR, Kalra M, Jeffries JL, Carroll JL, Bean JA, Witt SA, Glascock BJ, Daniels SR. Left ventricular function in children with sleep-disordered breathing. Am J Cardiol. 2005 Mar 15;95(6):801-4. doi: 10.1016/j.amjcard.2004.11.044. PMID 15757619
- [Background] Kalra M, Kimball TR, Daniels SR, LeMasters G, Willging PJ, Rutter M, Witt SA, Glascock BJ, Amin RS. Structural cardiac changes as a predictor of respiratory complications after adenotonsillectomy for obstructive breathing during sleep in children. Sleep Med. 2005 May;6(3):241-5. doi: 10.1016/j.sleep.2004.10.004. Epub 2004 Dec 10. PMID 15854854
- [Derived] Witter AM, Smith DF, Khan MTF, Nakamura A, Schuler CL, DiFrancesco MW, Hossain MM, Amin RS. Relationship of Circadian Blood Pressure Dysregulation With Left Ventricular Structure and Function in Children With Obstructive Sleep Apnea. J Sleep Res. 2025 Oct;34(5):e70049. doi: 10.1111/jsr.70049. Epub 2025 Apr 1. PMID 40170220
- [Derived] Domany KA, Huang G, Hossain MM, Schuler CL, Somers VK, Daniels SR, Amin R. Effect of Adenotonsillectomy on Cardiac Function in Children Age 5-13 Years With Obstructive Sleep Apnea. Am J Cardiol. 2021 Feb 15;141:120-126. doi: 10.1016/j.amjcard.2020.11.019. Epub 2020 Nov 19. PMID 33220319